CLINICAL TRIAL: NCT00624299
Title: Botulinum Toxin: an Adjunct in Limb Reconstruction - Can it Reduce Pain and Joint Complications in the Lengthening Phase?
Brief Title: Botox Clinical Trial
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: A similar study had already been conducted, therefore pursuing this trial would have been unethical
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Dr Jim Bonham, Sheffield Children's NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCH-07-006
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Leg Length Inequality; Foot Deformities
Keywords: botox; limb reconstructions; limb reconstruction surgery
MeSH Terms: conditions — Leg Length Inequality; Foot Deformities | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox (Experimental): Botox
  Interventions: Drug: Botox
- Placebo (Placebo Comparator): Saline injection
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Botox — Botox injection (100 ius) per muscle
  Arms: Botox
Other: Saline — Saline injection
  Arms: Placebo

SUMMARY:
The surgery to correct leg & foot deformities in children is a lengthy, & sometimes, difficult procedure. Metal frames are attached to the leg and / or foot and over a period of time the frame is manipulated to obtain the corrected position. During this period the muscles & skin become very tight which causes pain & may pull the joint out of position. When this happens it is sometimes necessary to stop the treatment before the best position is obtained. This means that not only is the child left with an inadequate result but that further surgery is required in the future.

If the tension could be removed whilst the treatment is underway this would reduce the pain, the possibility of joint damage & potentially allow a more satisfactory to be obtained without the need for further surgery.

Botulinum toxin or Botox, as it is commonly called, has the potential to temporarily reduce the tension in the muscles without causing permanent damage.

DETAILED DESCRIPTION:
Excessive soft tissue tension (i.e.. tight muscles and associated tissues) is the most limiting factor in lengthening and correction of limb length deficiency. Bone lengthening is achieved by surgically breaking the bone and with the use of an extending device, commonly placed on the outside of the limb, the bones ends are distracted. One millimetre a day is commonly the amount of distraction, however the soft tissue increases in length at a slower pace than the bone which leads to soft tissue tension.

Excessive soft tissue tension leads to:

* Soft tissue contractures temporary or permanent short muscles and tendons
* Joint subluxation or instability joints which slip out of line and are loose
* Pain
* Loss of function inability to move joints properly and difficulty walking This puts the joint in a very vulnerable situation and increases the possibility of subluxation. A similar problem arises during tibial lengthening, when the ankle takes up an equinus position (foot pointing down and in). Both deformities reduce the functional ability of the child and risk the joint becoming permanently damaged.

Increasing pain levels accompany these deformities leading to a greater reluctance to comply with treatment or rehabilitation. The lack of joint mobility has further detrimental effect on the limb as it becomes weak and stiff.

These events become a vicious cycle which is difficult to resolve without further intervention. When soft tissue tension is becoming a problem, i.e. pain levels are increasing and difficult to control, or the joint is under threat of instability, the first course of action is to slow or stop the lengthening for a few days which allows the soft tissue tension to decrease. The drawback with this is the potential for the bone ends to start fusing and prevent further lengthening once the process is resumed. To re start the process means the child has to have a further general anaesthetic to enable the bone to be re osteotomised (re broken).

Online Form 6 Some groups of children who undergo lengthening are more susceptible to soft tissue tension than others and therefore prophylactic surgical measures are employed. In anticipation of the soft tissue tension muscles known to create problems are commonly selected for surgical releases. This has been shown to be an effective method for reducing the effects of the tension but it is not without its problems. Releases done at the time of surgery may heal before the lengthening is complete and may need to be repeated. Releases cause trauma to the muscle or tendon which then heals by scar tissue, a structure known to be less pliable than specialised muscle or tendon tissue. Regaining long term function can be compromised.

Temporarily reducing soft tissue tension during the lengthening phase of treatment which has no long term consequences would be an ideal situation. Botulinum toxin has the ability to do this. Paley (2004) used Botulinum toxin as an adjunct to or in place of soft tissue release during femoral lengthening and noted that it seemed to reduce muscle spasm and pain in patients. Unfortunately this was not supported by any form of evaluative research.

ELIGIBILITY:
Inclusion Criteria:

* Any child with femoral, tibial deformity or CTEV having limb reconstruction surgery which involves the distraction of bone and or soft tissue.

Exclusion Criteria:

* Children with neurological aetiology

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
The pain levels using a visual analogue scale validated at the Sheffield Children's Hospital | 2 years

SECONDARY OUTCOMES:
Range of movement in affected joints measured by a goniometre | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria Burton, Principal Investigator — Sheffield Children's Hospital
Locations (1):
- Clinical Research Facility, Sheffield Children's Hospital, Sheffield, South Yorkshire, United Kingdom